CLINICAL TRIAL: NCT05367037
Title: Physiological Ventricular Pacing Versus Managed Ventricular Pacing for Persistent Atrial Fibrillation Prevention in Patients With Prolonged Atrioventricular Interval: a Multicenter RCT
Brief Title: Physiological Ventricular Pacing Vs Managed Ventricular Pacing for Persistent AF Prevention in Prolonged AV Interval
Acronym: PhysioVP-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quovadis Associazione (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PhysioVP-AF
Record Dates: First submitted 2022-01-12; First posted 2022-05-10 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Sinus Node Disease; Atrioventricular; Block, Second Degree (Types I and II)
Keywords: Sinus Node Disease; Paroxysmal AV-block; conduction system pacing; persistent atrial fibrillation
MeSH Terms: conditions — Sick Sinus Syndrome; Bites and Stings; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: a prospective, randomized study in a 1:1 ratio, single-blind with double-blind evaluation (the actual evaluator of the primary endpoint is the pacemaker device's internal diagnostic algorithm, without intervention by the Investigator)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: single-blind with double-blind evaluation (the actual evaluator of the primary endpoint is the pacemaker device's internal diagnostic algorithm, without intervention by the Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PhysioVP group (Active Comparator): Physiological ventricular pacing
  Interventions: Device: PhysioVP
- DDD-VPA group (Active Comparator): Dual-chamber pacing with the addition of algorithms for ventricular pacing avoidance
  Interventions: Device: DDD-VPA

INTERVENTIONS:
Device: PhysioVP — The Physiological ventricular pacing is achieved by delivering a stimulus to a cardiac conduction structure, such as the bundle of His or left bundle branch of the His-Purkinje system, with a permanent lead. PhysioVP activates the heart through the native His-Purkinje conduction system, thus offering the most physiologic pacing approach to correct the PR interval and avoiding pacing-induced dyssynchrony. A specialized delivery sheath for His-Purkinje system pacing with appropriate or standard leads will be used. The atrial leads will be implanted in the right atrial appendage and will connect the leads to the standard dual-chamber PM. By continuously recording a 12-lead ECG, we determine whether cardiac conduction structure, such as the bundle of His or left bundle branch of the His-Purkinje system, will be achieved.
  Arms: PhysioVP group
Device: DDD-VPA — In dual-chamber pacing with the addition of algorithms for ventricular pacing avoidance, also called managed ventricular pacing, the right ventricular (RV) lead is implanted in the myocardial right ventricular (septum or apex). In this pacing mode, the ventricular pacing is minimized by using algorithms for right ventricular pacing avoidance. Therefore, the RV leads will be implanted in the right ventricular myocardial sites (septum or apex) and standard bipolar active or passive fixation leads. In addition, the atrial leads will be implanted in the right atrial appendage and connect leads to the standard dual-chamber PM.
  Arms: DDD-VPA group

SUMMARY:
A multicenter, prospective, randomized study in a 1:1 ratio, single-blind with double-blind evaluation to evaluate the superiority of physiological ventricular pacing (proposed modality) vs. managed ventricular pacing (control) for prevention of persistent AF (PeAF) occurrence in patients with prolonged atrioventricular interval (PR≥180 ms) and indication for pacing: sinus node disease and/or paroxysmal type 1 or 2-second degree AV block.

DETAILED DESCRIPTION:
Study aim: Evaluate the superiority of physiological ventricular pacing (proposed modality) vs. managed ventricular pacing (control) for prevention of persistent AF (PeAF) occurrence in patients with prolonged atrioventricular interval (PR≥180 ms) and indication for pacing: sinus node disease and/or paroxysmal type 1 or 2-second degree AV block. If the efficacy superiority is confirmed, this pacing mode may be considered to reduce the occurrence of persistent atrial fibrillation in this group of patients.

Study design: Independent, multicenter, prospective, randomized study in a 1:1 ratio, single-blind with double-blind evaluation (the actual evaluator of the primary endpoint is the pacemaker device's internal diagnostic algorithm, without intervention by the Investigator). This study will use only CE-marked devices already part of clinical practice.

Groups:

* PhysioVP group: the Physiological Ventricular Pacing is achieved by delivering a pacing stimulus to a cardiac conduction structure, such as the bundle of His or left bundle branch of the His-Purkinje system, with a permanent lead. PhysioVP activates the heart through the native His-Purkinje conduction system, thus offering the most physiologic pacing approach to correct the PR interval and avoiding pacing-induced dyssynchrony.
* DDD-VPA group: In managed ventricular pacing, the right ventricular (RV) lead is implanted in the myocardial right ventricular (septum or apex). In this pacing mode, the ventricular pacing is minimized by using algorithms for right Ventricular Pacing Avoidance.

Devices used:

* PhysioVP group: a specialized delivery sheath for His-Purkinje system pacing with appropriate or standard leads will be used.
* DDD-VPA group: the RV leads will be implanted in the standard right ventricular myocardial sites (septum or apex) using standard bipolar active-fixation leads.

The atrial leads will be placed in the right atrial appendage in both groups. The 13 participating Italian Clinical Centers are proven experience in the PM implantation procedures used in the study.

Enrolled patients will be monitored by in-office clinical checks at 1, 12, 24, and 36 months and by home monitoring at 6, 18, and 30 months after implantation.

ELIGIBILITY:
Inclusion Criteria:

18 years older patients, able to express Informed Consent, with prolonged atrioventricular interval (PR>180 ms) and one of the following indications for PM implantation according to current guidelines:

* Sinus node disease.
* Paroxysmal type1or 2 second-degree AV-block.

Exclusion Criteria:

* Candidacy for implantable cardioverter-defibrillator or cardiac resynchronization therapy device implantation.
* Severe grade mitral or aortic regurgitation/stenosis.
* Atrial fibrillation ablation (left pulmonary veins).
* Cardiac surgery < 3 months before PM implantation.
* History of long-standing persistent AF.
* Permanent third-degree AV block.
* Participation in another clinical trial in the past 3 months.
* Pregnancy or intention to become pregnant.
* Life expectancy of < 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
PeAF Free | 36 months
  Freedom from persistent AF occurrences up to 36 months after the pacemaker (PM) implant.
  The occurrence of PeAF is defined as the first AF / Atrial Flutter / Atrial Tachycardia episode lasting > 7 days, detected by the PM after a 1-month post PM lead-stabilization period. A day of AF is satisfied with a device-detected daily AF burden of ≥ 23 hours. Device-detected AF may also be collected by remote monitoring tools, if available. The definition also includes the occurrence of episodes terminated by cardioversion, whatever its duration or undergoing AF ablation
Clinical composite outcome | 36 months
  Composite outcome based on the occurrence of one or more of the events: Death from cardiovascular disease, or heart failure, or pacing system upgrading to the conduction system pacing (CSP) or to the biventricular pacing (BVP).

SECONDARY OUTCOMES:
Hemodynamic performance, LV remodeling 1 | 12 months
  Echocardiographic parameters: Left Ventriculi end-systolic volume (ml/m2).
Hemodynamic performance, LV remodeling 2 | 12 months
  Echocardiographic parameters: LVEF (%).
Hemodynamic performance, Diastolic function 1 | 12 months
  Echocardiographic parameters: E to A mitral wave amplitude ratio.
Hemodynamic performance, Diastolic function 2 | 12 months
  Echocardiographic parameters: E wave deceleration time (ms).
Hemodynamic performance, Diastolic function 3 | 12 months
  Echocardiographic parameters: pulsed-wave tissue Doppler early diastolic septal mitral annular velocity (e') (cm/s).
Hemodynamic performance, Diastolic function 4 | 12 months
  Echocardiographic parameters: E/e' ratio.
Hemodynamic performance, Diastolic function 5 | 12 months
  Echocardiographic parameters: Diastolic time (from onset E wave to end A wave) normalized for RR interval (ms).
Hemodynamic performance, Left atrial volume | 12 months
  Echocardiographic parameters: Left atrial volume (ml/m2).
Hemodynamic performance, Mitral regurgitation | 12 months
  Echocardiographic parameters: vena contracta (mm).
Clinical evaluations, NYHA | 12, 24, and 36 months
  NYHA class variation (I, II, III, IV).
Clinical evaluations, MLHFQ | 12, 24, and 36 months
  Variation of Quality-of-Life assessment by Minnesota Living with Heart Failure questionnaire (MLHFQ).
Clinical evaluations | 12, 24, and 36 months
  Number of cardiovascular diseases related to health structure access.
Safety endpoints, PRAE | 36 months
  Rate of all procedure-related adverse events (PRAE).
Safety endpoints, Potentially harmful factor 1 | 36 months
  Implantation/s procedure time (mm:ss).
Safety endpoints, Potentially harmful factor 2 | 36 months
  Fluoroscopy time (mm:ss).
Safety endpoints, Incidence Rate of re-interventions | 36 months
  Rate of re-interventions for lead revision, replacement, or infection.
Estimated battery longevity | 36 months
  Estimated residual battery longevity (time to end-of-life) by the implanted device every 6-months and/or when the primary endpoint is reached.

CONTACTS AND LOCATIONS:
Overall Officials: Gianni Pastore, MD, Principal Investigator — Cardiology Unit, "S.Maria della Misericordia" Hospital, Rovigo, Italy
Locations (1):
- Elettrofisiologia, Cardiologia, Ospedale di Rovigo, Rovigo, Veneto, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pastore G, Bertini M, Bonanno C, Coluccia G, Dell'Era G, De Mattia L, Grieco D, Katsouras G, Maines M, Marcantoni L, Marinaccio L, Paglino G, Palmisano P, Ziacchi M, Zoppo F, Noventa F. The PhysioVP-AF study, a randomized controlled trial to assess the clinical benefit of physiological ventricular pacing vs. managed ventricular pacing for persistent atrial fibrillation prevention in patients with prolonged atrioventricular conduction: design and rationale. Europace. 2023 May 19;25(5):euad082. doi: 10.1093/europace/euad082. PMID 36974970
- See also: Promotor's site — https://www.quovadis-ass.it/physiovp-af-trial/